CLINICAL TRIAL: NCT03232632
Title: Assessment of Cardiac Fixation During Positron Emission Tomography (PET) Examination Using 18F-Flutemetamol (Vizamyl ®) Within Amyloid Cardiac Injuries.
Brief Title: Assessment of Cardiac Fixation During PET Using a New Drug Within Amyloid Cardiac Injuries.
Acronym: AMYLCAR
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: intervention programming
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13 199 02
Record Dates: First submitted 2017-01-11; First posted 2017-07-28 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; flutemetamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET with 18 F-Flutemetamol (Experimental): PET with 18 F-Flutemetamol (Vizamyl®) = product under Alzheimer's disease indication
  Interventions: Drug: PET with 18 F-Flutemetamol

INTERVENTIONS:
Drug: PET with 18 F-Flutemetamol — PET with 18 F-Flutemetamol (Vizamyl ®)
  Other Names: Vizamyl®

SUMMARY:
To estimate distribution's parameters of 18F-Flutemetamol (Vizamyl®) fixation on myocardium for patients with amyloid cardiac injuries.

DETAILED DESCRIPTION:
Hypothesis had been performed that PET with 18F-Flutemetamol (Vizamyl®) could lead an early diagnostic. Indeed, this tracer had been recently used to highlight inter-cerebral beta-amyloid plaques on patients with Alzheimer Disease.

Because this labelling is performed on amyloid deposits, this tracer would lead to view and to quantify amyloid deposits within cardiac amyloid injuries.

Results of this PET will be combined with scan examinations for a better anatomic tracking.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed for amyloidosis with proved cardiac injury or strongly suspected:

  * cardiac echography with typical signs of amyloid injury,
  * anatomical result confirming presence of amyloid deposits at cardiac or peripheral level
* Signature of Informed Consent Form,
* Affiliation to a social security system

Exclusion Criteria:

* Patient who suffers from another pathology which could lead cardiac injury (coronary disease, valvular disease, other pathology of deposit),
* Pregnancy and lactating women,
* Absence of effective contraception,
* Irradiating examination performed within the last 12 months or scheduled within the next 12 months,
* Unable patient physically, mentally or legally to provide informed consent,
* Patient under a system of legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
ratio Heart/ Upper Mediastinum | average of last 15 minutes
  peak of 18F-Flutemetamol capture
standardized uptake value (SUV) measures | average of last 15 minutes
  standardized uptake value (SUV) measures

CONTACTS AND LOCATIONS:
Overall Officials: Eric OUHAYOUN, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No